CLINICAL TRIAL: NCT00119483
Title: Older Men and Testosterone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Eldre menn og testosteron
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Hypogonadism
Keywords: Men; testosterone; hypogonadal; aging; body composition; quality og life; Muscle strength; Aging male
MeSH Terms: conditions — Hypogonadism; Multiple Endocrine Neoplasia Type 1 | interventions — testosterone undecanoate

INTERVENTIONS:
Drug: Nebido (Testosterone Undecanoate)

SUMMARY:
Male hypogonadism is a clinical situation characterized by a low serum testosterone level in combination with a diversity of symptoms and signs such as reduced libido and vitality, decreased muscle mass, increased fat mass and depression. Similar symptoms in combination with subnormal testosterone levels are seen in some elderly men. Low testosterone levels are associated with known cardiovascular risk factors, and men with diabetes and stroke have lower testosterone levels than healthy men. Even though several publications have suggested that testosterone treatment in hypogonadal men may have beneficial effects, it is still uncertain if testosterone substitution in the aging man is indicated. Despite this uncertainty the sale of testosterone has increased enormously the last few years.

We hypothesize that older men with subnormal testosterone levels have a varying degree of dysfunction/symptoms both physically and mentally, and that these dysfunction/symptoms can be improved with testosterone treatment.

DETAILED DESCRIPTION:
Older men and testosterone (Short version of the study protocol)

Cohort study "How is life as an elderly man when serum testosterone is subnormal?"

To investigate whether subnormal testosterone levels in elderly men (60-80 years old) is associated with clinical symptoms and/or disease, the investigators will ask men with normal testosterone (>11.3 nmol/l) and men with subnormal testosterone levels (<11.3 nmol/l) who participated in the last Tromsø study 2001 to participate in this study.

Screening: Blood pressure, clinical examination including prostate examination, blood samples (testosterone, SHBG, LH, FSH, albumin and PSA).

Aproximately 350 men had subnormal testosterone levels in the last Tromsø study and the researchers will try to include up to 200 men who still have subnormal testosterone levels and up to 200 age matched men who still have normal testosterone levels.

Procedures

Symptoms: Aging Male Symptom Score

Muscle strength and function: The researchers will investigate muscle strength, peak torque with isokinetic dynamometry in the knee joint and muscle function (gait, balance and movement); Grip Strength

Neuropsychological tests

* Cognitive function level: WAIS
* Memory: Wechslers Memory Scale Revised (WMS-R)
* Trail making A and B.
* Attention and concentration: Knox cube
* Cognitive flexibility: Word fluency test and Stroop test
* Quality of life: GHQ - 30 with Likert score
* Depression: Beck Depression Inventory

The metabolic syndrome

* DEXA (Lunar Prodigy): *Whole body, body composition; *Lumbar spine and hip, bone mineral density
* CT scan of the abdomen to distinguish intra vs. subcutaneous fat deposits.
* Oral glucose tolerance test.
* Lipid profile /per oral fat load. (80 men will take part in this investigation)
* Examination of the androgen receptor, especially the CAG and GGN polymorphism of the androgen receptor has been associated with glucose and fat metabolism.
* Blood pressure and heart rate.
* Neuroendocrine regulation: LH, FSH, SHBG, estradiol, testosterone, cortisol, ACTH, IGF-1, IGFBP-3, TSH, FT4, prolactin and leptin.
* Sleep

Interventions study "Should subnormal testosterone levels be treated?"

To investigate whether older men with subnormal testosterone levels would benefit from physiological testosterone supplementation, the men with subnormal testosterone levels participating in the cohort study (approximately 150-200 men) will be asked to participate in a one year intervention study.

Randomization and treatment:

Double blind randomized (1:1) 1-year study. First injection at inclusion, second after 6 weeks, the third injection after 16 weeks, the fourth at 28 weeks and the last at 40 weeks. Active treatment is Nebido, 1000 mg testosteron undecanoate, a 4 ml intramuscular depot injection. Schering AS will supply the study with both Nebido and placebo (containing "castor oil" and "benzyl benzoate").

Registration of adverse events:

All adverse events will be recorded in the participants CRF. Serious adverse events will be reported according to regulations.

Procedures:

The above-described procedures for the cohort study will also be performed in the intervention study.

Testosterone levels, hematocrit, creatinine, ALAT and PSA will be controlled at every visit.

Object variables for both the cohort and intervention study

Primary:

Psychosexual quality of life; Muscle strength

Secondary:

Muscle function; Body composition; Intraabdominal vs. subcutaneous fat distribution; CAG and GGN polymorphism in the androgen receptor gene; Bone mineral density; Per oral glucose tolerance test; Lipid profile/fat tolerance test; Neuropsychological test; Neuroendocrine regulation Sleep

Statistics and methods:

The study will be performed at the Clinical research ward at the University Hospital of North Norway.

Comparisons between the groups will be assessed with non-parametrical tests (Mann-Whitney U-test) or ANOVA with a significant level p<0.05. In the intervention study delta-values will be used to assess changes during treatment and differences between the study groups. SPSS will be used as statistical program.

Inclusion of patients to the cohort study should be completed during 2006 and the intervention study should be completed during 2007.

Research partner Johan Svartberg, Department of Medicine, University Hospital of North Norway, Tromsø, Norway is the responsible investigator.

Partners: Professor Rolf Jorde and John-Bjarne Hansen MD, PhD, Department of Medicine, Professor Johan Sundsfjord, Department of Clinical Chemistry and Professor Knut Waterloo, Department of Neurology, University Hospital of North Norway, Tromsø, Norway and Professor Aleksander Giwercman, Scanian Andrology Center, Department of Urology, Malmö University Hospital, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Men 60-80 years old
* Serum-testosterone levels <11.0 nmol/l
* Signed informed consent.

Exclusion Criteria:

* Prostate cancer
* Breast cancer
* Liver tumor/cancer
* Unstable angina
* Untreated congestive heart disease
* Epilepsy
* Migraine
* Hematocrit >50%
* PSA >4.0 ug/l
* Serum creatinine >130 umol/l
* ALAT >100 U/l
* Known intolerance to testosterone undecanoate
* Participation in another research trial.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Quality of life (psycho-sexual)
Muscle strength

SECONDARY OUTCOMES:
Body composition
Muscle function
Intra abdominal vs subcutanous fat mass.
Bone density
CAG and GGN polymorphy in the androgene receptor gene
Glucose tolerance/insulin resistance
Fat tolerance
Neuroendocrine profile
Neuropsychological profile
Sleep

CONTACTS AND LOCATIONS:
Overall Officials: Johan Svartberg, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- Department of Medicine, University Hospital of North Norway, Tromsø, Norway